CLINICAL TRIAL: NCT01152112
Title: A Hysteroscopic Office Myomectomy Evaluation Using the MyoSure Tissue Removal System for the Removal of Uterine Fibroids and Polyps in the Treatment of Abnormal Uterine Bleeding (AUB)
Brief Title: HOME Study: Hysteroscopic Office Myomectomy Evaluation
Acronym: HOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hologic, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMP 2009003
Record Dates: First submitted 2010-06-18; First posted 2010-06-29 (Estimated); Results first posted 2017-09-13 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-08

CONDITIONS: Uterine Fibroids; Polyps
Keywords: morcellator; hysteroscope; myomectomy; polypectomy; uterine fibroids; uterine polyps; office; cost; local anesthetic; cervical block; pain management
MeSH Terms: conditions — Leiomyoma; Polyps; Agnosia | interventions — Uterine Myomectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment, Office Setting, myomectomy (Experimental): Myomectomy for uterine polyps and/or fibroids occurring in an office setting
  Interventions: Device: Myomectomy
- Treatment, Hospital Setting, myomectomy (Experimental): Myomectomy for uterine polyps and/or fibroids occurring in a hospital setting
  Interventions: Device: Myomectomy

INTERVENTIONS:
Device: Myomectomy — Removal of fibroids and / or polyps
  Other Names: Fibroid removal; Polyp removal

SUMMARY:
The purpose of this study is to demonstrate safety and effectiveness of the MyoSure Tissue Removal System when used by community gynecologists in an office setting for the treatment of patients with symptomatic intrauterine polyps and submucosal fibroids.

DETAILED DESCRIPTION:
Approximately one hundred subjects will be enrolled in a randomized, comparative setting study conducted at 10-15 investigational sites. Sixty subjects will be randomized to undergo treatment in an office setting, and 40 subjects will be randomized to undergo treatment in a hospital or ambulatory surgical center (ASC) setting. Subjects will undergo a hysteroscopic tissue removal procedure to remove intrauterine polyps, type 0 fibroids, or type I fibroids. Saline infused sonohysterogram images (SIS) obtained at three months post treatment will be compared to pre-treatment images, to determine the percent reduction in target pathology volume. Additionally, subject self-reported pain scores (as rated on an 11 point scale) will compare pain occurring during the treatment procedure to the average pain level experienced during a PAP smear. Economic data will be collected and compared between the two treatment settings.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female between 18 and 55 years of age
* Subject must be able to understand, read and sign the study specific informed consent forms after the nature of the study has been fully explained to her
* Subject is a pre-menopausal or peri-menopausal female, either nulliparous or parous
* Subject is experiencing AUB as confirmed by a symptom raw score of 23 or a calculated symptom score of 44.0 or higher on the Uterine Fibroid Scale and Health Related Quality of Life (UFS-QOL)
* Subject is indicated for myomectomy or polypectomy for benign appearing pathology, based on a hysteroscopic exam and measured by saline infused sonogram assessment within 30 days of the planned index procedure
* Subject exhibits intrauterine polyps and/or submucous myomas which, in the opinion of the treating physician, are compatible with office-based treatment (e.g. 15 minutes or less of cutting time) using the MyoSure device and meet at least one of the following criteria:
* One or more polyps, with at least one of the polyps ≥ 1.5 cm and ≤ 3.0 cm diameter and having broad based attachment to the uterine wall.
* Up to two Type 0 or Type 1 myomas with at least one of the myomas being ≥ 1.5 cm and none of the myomas being 3.0 cm diameter

  * If the first myoma is 3.0 cm, the second myoma must be ≤ 2.0 cm
  * Fundal myomas must be Type 0
* Polyps plus up to two Type 0 or Type I myomas with at least one of the myomas being ≥ 1.5cm and ≤ 3.0 cm
* The subject demonstrates a negative pregnancy test within 48 hours prior to the planned index procedure
* The subject must document a score of 5 or lower on the Pap Smear and Blood Draw scales of the Pain Tolerance Survey

Exclusion Criteria:

* Subject has known or suspected cancer, including breast, endometrial, and ovarian
* Contraindication and/or allergy to local anesthetic, or oral medications specified in the treatment protocol
* The subject has a history of chronic narcotic use
* Previous uterine artery embolization or other uterine artery occlusion procedure (Doppler or laparoscopic)
* Subject has blood borne pathogens-HIV, hepatitis B, CJD, etc.
* Subject has an IUD at the time of the procedure. A subject may be enrolled in the study if the IUD is removed prior to the treatment procedure
* Subject is taking an anticoagulant or antiplatelet medication other than low dose aspirin
* Active pelvic inflammatory disease or pelvic/vaginal infection
* Subject has a known or suspected coagulopathy or bleeding disorder
* Subject has a history of unmanaged endocrine disease
* Subject has current or past, acute or chronic psychiatric disorder which, in the opinion of the Investigator, may preclude proper evaluation and follow-up
* Subject has a history of auto-immune, inflammatory, or connective tissue disease
* Subject has a history of disease which increases the risk for fluid overload (i.e. significant cardiac, hepatic, or renal dysfunction)
* Uncontrolled hypertension lasting two years or more
* Use of any experimental drug or device within 30 days prior to the screening visit
* The subject has a terminal illness that may prevent the completion of any follow-up assessments
* Any employee or relative of an employee of the Sponsor company or any Investigator site employee or relative of employees working on the study
* Subject has other co-morbid condition(s) that, in the opinion of the Investigator, could limit the subject's ability to participate in the study or impact the scientific integrity of the study
* Subject has one of the following:

  * Type II submucosal myoma
  * Type O or Type I submucosal myoma > 3.0 cm
  * Fundal Type I myoma
  * Highly vascularized myoma as determined by SIS or hysteroscopic examination

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2010-06; Primary Completion 2012-01 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Evantash, MD, Study Director — Sponsor GmbH
Locations (9):
- United States (9):
  - Phoenix Gynecology Consultants, Phoenix, Arizona
  - Boulder Women's Clinic, Boulder, Colorado
  - Women's Health Care Practice, Champaign, Illinois
  - The Research Division for Integrated Health Services, Ann Arbor, Michigan
  - Rubino OB/Gyn, West Orange, New Jersey
  - Williams, Benavides, Marston, & Kaminski, Raleigh, North Carolina
  - Complete Healthcare for Women, Columbus, Ohio
  - Kulbresh Women's Center, Irmo, South Carolina
  - Obstetrics and Gynecology, North Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
The Journal of Minimally Invasive Gynecology

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment, Office Setting, Myomectomy | Treatment, Hospital Setting, Myomectomy
Started | 42 | 32
Completed | 42 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment, Office Setting, Myomectomy | Treatment, Hospital Setting, Myomectomy | Total
Number analyzed (Participants) | 42 | 32 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 32 | 74
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 32 | 74
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 42 | 32 | 74

OUTCOME MEASURES:

1. Primary Outcome: Percent Reduction in Target Pathology Volume
Description: Percent reduction in target pathology volume, compared between pre-treatment baseline and 3 months post MyoSure treatment
Time Frame: Three months post treatment
Population: A total of 108 pathologies were removed in 74 patients. Among the 108 pathologies removed, 53 were removed in the office setting (28 myomas, 25 polyps) and 55 were removed in the ASC setting (14 myomas, 41 polyps).
Measure: Mean (95% Confidence Interval); unit: percentage of fibriods/polyps
Units Other Than Participants: Fibroids and Polyps
Arm/Group | Treatment, Office Setting, Myomectomy | Treatment, Hospital Setting, Myomectomy
Number analyzed (Participants) | 42 | 32
Number analyzed (Fibroids and Polyps) | 53 | 55
percentage of fibriods/polyps | 96.9 [90.3 to 103.5] | 99.9 [99.6 to 100.2]

2. Secondary Outcome: Percent of Subjects That Achieve 100% Removal of Target Pathology
Description: Percent volume reduction of target pathology between baseline and month three post treatment assessments, as measured by saline infused sonohysterogram.
Time Frame: Three months post treatment
Reporting Status: Not Posted

3. Secondary Outcome: Subject Self-reported Pain Score Occurring During the Treatment Procedure
Description: Mean difference in pain score compared between subject-rated assessment of pain occurring during a pap smear and pain occurring during the MyoSure treatment procedure, based on the Wong-Baker Faces Rating Scale (FRS)
Time Frame: 1 hour post treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse effect information was collected throughout the study. All adverse effects were monitored until they were adequately resolved or explained.
Arm/Group | Treatment, Office Setting, Myomectomy | Treatment, Hospital Setting, Myomectomy
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/32
Other Adverse Events (participants affected / at risk) | 1/42 | 2/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment, Office Setting, Myomectomy (N=42) | Treatment, Hospital Setting, Myomectomy (N=32)
Food Poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) — Food Poisoning
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) — Food Poisoning
Pain (General disorders) | 1 (1) | 0 (0) — Pain and discomfort NEC

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No